CLINICAL TRIAL: NCT05125016
Title: Phase 1/2 Study of REGN4336 (a PSMAxCD3 Bispecific Antibody) Administered Alone or in Combination With Cemiplimab or REGN5678 (a PSMAxCD28 Bispecific Antibody) in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Trial to Find Out if REGN4336 is Safe and How Well it Works Alone and in Combination With Cemiplimab or REGN5678 for Adult Participants With Advanced Prostate Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R4336-ONC-20104; 2022-502130-17-00 (Other: EUCT Number)
Record Dates: First submitted 2021-10-25; First posted 2021-11-18 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Treatment-experienced metastatic castration-resistant prostate cancer (mCRPC)
MeSH Terms: interventions — cemiplimab; sarilumab

STUDY DESIGN:
Intervention Model Description: The study contains 3 separate modules in parallel: monotherapy with REGN4336 (Module 1) and combination therapies: REGN4336 plus cemiplimab (Module 2) and REGN4336 plus REGN5678 (Module 3). All 3 modules contain independent dose escalation cohorts and up to 2 recommended phase 2 dose regimens during dose expansion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Module 1- Monotherapy (Experimental): REGN4336
  Interventions: Drug: REGN4336; Drug: Sarilumab
- Module 2-Combo Therapy (Experimental): REGN4336 + Cemiplimab
  Interventions: Drug: REGN4336; Drug: Cemiplimab; Drug: Sarilumab
- Module 3-Combo Therapy (Experimental): REGN4336 + REGN5678
  Interventions: Drug: REGN4336; Drug: REGN5678; Drug: Sarilumab

INTERVENTIONS:
Drug: REGN4336 — Administered once weekly (QW) by subcutaneous (SC) injection, or intravenous (IV) infusion
Drug: Cemiplimab — Administered concomitantly every 3 weeks (Q3W) by IV infusion
  Other Names: REGN2810
  Arms: Module 2-Combo Therapy
Drug: REGN5678 — Administered concomitantly QW by IV infusion
  Arms: Module 3-Combo Therapy
Drug: Sarilumab — Administered once by IV infusion as prophylaxis prior to REGN4336 IV
  Other Names: REGN88; SAR153191

SUMMARY:
This study is researching an investigational drug called REGN4336. Some participants may receive additional investigational drugs in combination with REGN4336. These additional drugs include REGN5678, cemiplimab and sarilumab.

The main purpose of this study is to determine the safety, tolerability (how the body reacts to the drug) and effectiveness of REGN4336 alone, in combination with cemiplimab, or in combination with REGN5678. REGN4336, cemiplimab and REGN5678 are a type of treatment for cancer called immunotherapy,and are intended to activate T-cells to attack cancer cells.

This study has 2 parts. The purpose of Part 1 is to determine a safe dose of REGN4336 when given alone or when given in combination with cemiplimab or REGN5678. The purpose of Part 2 is to use the REGN4336 dose(s) determined in Part 1 to further test how well REGN4336 works to shrink tumors either when given alone or in combination with cemiplimab or REGN5678.

This study is looking at several other research questions, including:

* What side effects may happen from taking REGN4336 alone, in combination with cemiplimab, or in combination with REGN5678?
* How much REGN4336 is in the blood at different times when it is given alone, in combination with cemiplimab, or in combination with REGN5678?
* Does the body make antibodies against the study drugs (REGN4336, cemiplimab, or REGN5678)?

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma of the prostate without pure small cell carcinoma
2. Metastatic, castration-resistant prostate cancer (mCRPC) with PSA value at screening ≥4 ng/mL that has progressed within 6 months prior to screening, according to 1 of the following:

   1. PSA progression as defined by a rising PSA level confirmed with an interval of ≥1 week between each assessment
   2. Radiographic disease progression in soft tissue based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria with or without PSA progression
   3. Radiographic disease progression in bone defined as the appearance of 2 or more new bone lesions on bone scan with or without PSA progression NOTE: Measurable disease per RECIST version 1.1 per local reading at screening is not an eligibility criterion for enrollment
3. Has progressed upon or intolerant to ≥2 lines prior systemic therapy approved in the metastatic and/or castration-resistant setting (in addition to androgen deprivation therapy [ADT]) including at least one second-generation anti-androgen therapy (e.g. abiraterone, enzalutamide, apalutamide, or darolutamide)

Key Exclusion Criteria:

1. Has received treatment with an approved systemic therapy within 3 weeks of dosing or has not yet recovered (ie, grade ≤1 or baseline) from any acute toxicities
2. Has received any previous systemic biologic or immune-modulating therapy (except for Sipuleucel-T) within 5 half-lives of first dose of study therapy, as described in the protocol
3. Has received prior PSMA-targeting therapy. Exception: Prior therapy with approved PSMA-targeted radioligand(s) is permitted
4. Any condition that requires ongoing/continuous corticosteroid therapy (>10 mg prednisone/day or anti-inflammatory equivalent) within 1 week prior to the first dose of study therapy
5. Ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments
6. Encephalitis, meningitis, neurodegenerative disease (with the exception of mild dementia that does not interfere with activities of daily living [ADLs]) or uncontrolled seizures in the year prior to first dose of study therapy
7. Uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection; or diagnosis of immunodeficiency, as described in the protocol.

NOTE: Other protocol defined Inclusion/Exclusion Criteria apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2027-01-14 (Estimated); Study Completion 2027-01-14 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | 28 days, up to 42 days
  Dose escalation
Incidence and severity of treatment-emergent adverse events (TEAEs) | Up to 5 years
  Dose escalation
Incidence and severity of Immune-mediated Adverse Events (imAEs) | Up to 5 years
  Dose escalation
Incidence and severity of Serious Adverse Events (SAEs) | Up to 5 years
  Dose escalation
Incidence and severity of adverse event of special interest (AESIs) | Up to 5 years
  Dose escalation
Number of patients with grade ≥3 laboratory abnormalities | Up to 5 years
  Dose escalation
REGN4336 monotherapy concentrations in serum | Up to 5 years
  Dose escalation
REGN4336 concentrations in serum in combination with cemiplimab | Up to 5 years
  Dose escalation
REGN4336 concentrations in serum in combination with REGN5678 | Up to 5 years
  Dose escalation
Objective response rate (ORR) per modified per modified Prostate Cancer Working Group 3 (PCWG3) criteria | Up to 5 years
  Dose expansion

SECONDARY OUTCOMES:
ORR per modified per modified PCWG3 criteria | Up to 5 years
  Dose Escalation
Incidence and severity of TEAEs | Up to 5 years
  Dose expansion
Incidence and severity of imAEs | Up to 5 years
  Dose expansion
Incidence and severity of SAEs | Up to 5 years
  Dose expansion
Incidence and severity of AESIs | Up to 5 years
  Dose expansion
Number of patients with grade ≥3 laboratory abnormalities | Up to 5 years
  Dose expansion
REGN4336 monotherapy concentrations in serum | Up to 5 years
  Dose expansion
REGN4336 concentrations in serum in combination with cemiplimab | Up to 5 years
  Dose expansion
REGN4336 concentrations in serum in combination with REGN5678 | Up to 5 years
  Dose expansion
Percentage of patients with ≥50% reduction in prostate specific antigen (PSA) from baseline, confirmed by a second PSA test ≥3 weeks later | Up to 5 years
  Dose escalation and expansion
Percentage of patients with ≥90% reduction in PSA from baseline, confirmed by a second PSA test ≥3 weeks later | UP to 5 years
  Dose escalation and expansion
Anti-drug antibodies (ADA) to REGN4336 | Up to 5 years
  Module 1
ADA to REGN4336 and cemiplimab | Up to 5 years
  Module 2
ADA to REGN4336 and REGN5678 | Up to 5 years
  Module 3

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (12):
- United States (12):
  - Stanford University Medical Center - Blake Wilbur Drive, Palo Alto, California
  - Norton Cancer Institute, Louisville, Kentucky
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Atrium Health Levine Cancer Institute, Charlotte, North Carolina
  - The Ohio State University James Cancer Hospital, Columbus, Ohio
  - Penn Medicine University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/